CLINICAL TRIAL: NCT04345822
Title: Effect of Cervical Compressive Myelopathy on the Autonomic Nervous System and Clinical Implication
Brief Title: Cervical Cord Compression and Hypertension
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Taipei Veterans General Hospital, Taiwan (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2019_12_003CC
Record Dates: First submitted 2020-03-31; First posted 2020-04-14 (Actual); Last update posted 2020-04-14 (Actual); Status verified 2020-04

CONDITIONS: Hypertension
Keywords: heart rate variability; cervical myelopathy; blood pressure; decompression
MeSH Terms: conditions — Hypertension | interventions — Laminectomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- normotension: patients without diagnosis or treatment for hypertension
  Interventions: Procedure: Decompression surgery
- hypertension: patients with diagnosis or treatment for hypertension
  Interventions: Procedure: Decompression surgery

INTERVENTIONS:
Procedure: Decompression surgery — The surgeries aim to relieve the myelopathy from cord compression
  Other Names: cervical spine decompression surgery

SUMMARY:
Myelopathy from cervical cord compression may induce hypertension and sympathetic hyperactivity. Anesthesia may suppress sympathetic activity and lead to hypotension that require vasopressor treatment. We aim to elucidate the causative factors for severe hypotension during anesthesia by prospective observational study.

DETAILED DESCRIPTION:
It had been reported the cervical spondylotic myelopathy may lead to the development of hypertension. Decompression surgeries ameliorated neurological symptoms as well as the blood pressure. The cause may be the abnormality of autonomic dysfunction developed after myelopathy. However, the evidence was weak. We have noticed a tendency of hypotension during anesthesia in patients undergroing cervical spine surgeries, especially in surgeries of long levels and hypertensive patients. Thus we postulate the autonomic activity is abnormal in patients with cervical myelopathy. Sympathetic hyperactivity developed in order to maintain adequate perfusion to the cervical cord. When patients are under anesthesia, the sympathetic tone is suppressed, thus leading to severe hypotension that require the treatment of inotropic treatment. Heart rate variability (HRV) is a good index of autonomic activity. Thus we plan to Therefore we will measure the HRV (analysis of ECG) and baroreflex activity (analysis of arterial line during the anesthesia) in patients undergoing cervical spine surgeries for decompression of cord compression perioperatively. The primary end-point is the comparison of severity of cord compression between normotensive and hypertensive patients with cervical myelopathy. The secondary end-point is to compare blood pressure and HRV pre- and postoperatively. The third end-point is to elucidate the causative factors for severe hypotension during anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* cervical spine surgery for cord compression

Exclusion Criteria:

* spinal cord injury
* ASA class >3
* chronic kidney disease
* congestive heart failure
* BMI>30
* atrial fibrillation/ flutter
* obstructive sleep apnea

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: We exclude patients with other cormobidity that might lead to hypertension or hypetension. we perfrom age and gender matched pair.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-02-01 (Actual); Primary Completion 2021-03-31 (Estimated); Study Completion 2021-08-31 (Estimated)

PRIMARY OUTCOMES:
change of blood pressure | one day before surgery, during surgery, 3 months after surgery, 6 months after surgery
  noninvasive blood pressure
change of hear rate variability | one day before surgery, during surgery, 3 months after surgery, 6 months after surgery
  from analysis of ECG
baroreflex activity | during surgery (anesthesia)
  from analysis of arterial blood pressure waveform

SECONDARY OUTCOMES:
change of Japanese Orthopaedic Association Scores | one day before surgery, 3 months after surgery, 6 months after surgery
  17 points neurological assessment for cervical spine pathology (from 0~17; 0 denotes worst neurological condition, 17 denotes intact )
change of the Nurick scores | one day before surgery, 3 months after surgery, 6 months after surgery
  6 grades neurological assessment for cervical spine pathology (Grade 0: no root or cord symptoms; 1, signs or symptoms of root involvement only; 2, signs of spinal cord involvement (normal gait); 3, mild gait abnormality (does not prevent employment); 4, gait abnormality prevents employment; 5, only able to walk with assistance; 6, chair bound or bedridden)

CONTACTS AND LOCATIONS:
Overall Officials: MC HO, MD, PhD, Study Chair — Taipei Veterans General Hospital, Taiwan
Locations (1):
- Taipei Veterans General Hospital, Taipei County, Taiwan